CLINICAL TRIAL: NCT05774496
Title: Pregnancy and Congenital Toxoplasmosis : Maternal and Child Risks Assessment, Data From Patients Followed-up in the Lyon Cohort
Brief Title: Pregnancy and Congenital Toxoplasmosis
Acronym: GRETA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_1041; 2022-A02496-37 (Other: ID-RCB)
Record Dates: First submitted 2023-02-16; First posted 2023-03-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Congenital Toxoplasmosis; Retinochoroiditis
MeSH Terms: conditions — Toxoplasmosis, Congenital; Chorioretinitis | interventions — Postpartum Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Congenital toxoplasmosis women: Women older than 21 suffering from congenital toxoplasmosis, with or without children.
  Interventions: Other: Estimation of the occurrence of retinochoroiditis in women with congenital toxoplasmosis and previous retinochoroiditis lesions (recurrence) during pregnancy and postpartum.

INTERVENTIONS:
Other: Estimation of the occurrence of retinochoroiditis in women with congenital toxoplasmosis and previous retinochoroiditis lesions (recurrence) during pregnancy and postpartum. — All fundus examinations completed during pregnancy and postpartum in women with congenital toxoplasmosis and previous retinochoroiditis lesions are going to be checked.

SUMMARY:
The Toxoplasma gondii parasite causes toxoplasmosis. It is characterized by persistent cysts mostly localised in the brain and ocular areas. In the case of immunodeficiency, those cysts are likely to reactivate. During pregnancy, an infection exposes the foetus to a variety of consequences, from severe neurologic lesions to subclinical forms at birth. However, those forms are likely to complicate at any age to toxoplasmic retinochoroiditis, that can unpredictably recur with severe functional consequences. Pregnancy may stimulate lesions or their recurrences, putting the foetus at risk of contamination because of the release of tachyzoites in the bloodstream. The occurrence of these complications is poorly known, especially with congenital toxoplasmosis. Nevertheless, this information is essential to take care of patients, particularly women with congenital toxoplasmosis, usually worried about the consequences of a pregnancy.

As a precaution, women with congenital toxoplasmosis follow a specific ophthalmologic, and trimonthly monitoring, composed of fundus examinations during pregnancy and in postpartum. To eliminate the contamination risk, serological examinations at birth and one year later are done on their kids.

The aim of this study is to estimate the risk of toxoplasmic retinochoroiditis during pregnancy and the impact on their children. Retrospective and prospective data from the Lyon Cohort of Maternal and Congenital Toxoplasma Infections will be used.

As a result of to this study, the investigators expect to provide better information to women suffering from congenital toxoplasmosis about their own ocular safety during pregnancy, and the safety of their child(ren). The investigators seek to provide new national and international recommendations about these patients and their children's care.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman
* Born before March 2022
* Suffering from congenital toxoplamosis

Exclusion Criteria:

* Refusal to give informed consent
* Any condition that would limit the ability of the patient to give consent
* Psychiatric cares
* To be deprived of liberty
* To be under administrative supervision

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The Lyon cohort is composed of 193 women suffering from a congenital toxoplasmosis confirmed at their birth in the parasitology and mycology unit of the La Croix-Rousse hospital, and they have been tracked since then.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-03-16 (Actual)

PRIMARY OUTCOMES:
The number of toxoplasmic retinochoroiditis during pregnancy in women with congenital toxoplasmosis and previous retinochoroiditis lesions (recurrence). | Toxoplasmic retinochoroiditis that occured during pregnancy (up to 40 weeks)
  All fundus examinations completed during pregnancy in women with congenital toxoplasmosis and previous retinochoroiditis lesions are going to be checked. The occurrence of retinochoroiditis during pregnancy will be compared to the occurrence of toxoplasmic retinochoroiditis during periods without pregnancy.
The number of toxoplasmic retinochoroiditis during postpartum in women with congenital toxoplasmosis and previous retinochoroiditis lesions (recurrence). | Toxoplasmic retinochoroiditis that occured during postpartum (up to 6 months after the delivery)
  All fundus examinations completed during postpartum in women with congenital toxoplasmosis and previous retinochoroiditis lesions are going to be checked. The occurrence of retinochoroiditis during postpartum will be compared to the occurrence of toxoplasmic retinochoroiditis during periods without pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Wallon, Principal Investigator — Service de parasitologie et mycologie médicale de l'Hôpital de la Croix-Rousse
Locations (1):
- Service de parasitologie et mycologie médicale, Lyon, France